CLINICAL TRIAL: NCT03318666
Title: A Pilot Randomized Controlled Trial of SOVA (Supporting Our Valued Adolescents), a Social Media Intervention for Adolescents With Depression and Anxiety and Their Parents to Increase Use of Mental Health Services
Brief Title: Supporting Our Valued Adolescents Pilot Randomized Controlled Trial
Acronym: SOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ana Radovic, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PRO17070601; 1K23MH111922-01A1 (NIH)
Record Dates: First submitted 2017-10-13; First posted 2017-10-24 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Depression; Anxiety
Keywords: Adolescent; Adolescent Medicine; Mental Health Services; eHealth; Online systems; Primary Health Care; Social media; Social support
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (EUC) (Active Comparator): Both arms will receive this intervention
  Interventions: Other: Enhanced Usual Care
- Supporting Our Valued Adolescents (SOVA) (Experimental): This arm will receive the SOVA intervention in addition to Enhanced Usual Care
  Interventions: Behavioral: Supporting Our Valued Adolescents (SOVA); Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Supporting Our Valued Adolescents (SOVA) — The SOVA intervention includes:
  * a welcome email to the websites (adolescents also get a SOVA intro video and mobile app)
  * adolescents will have access to the website specifically for adolescents: sova.pitt.edu
  * parents will have access to the website specifically for parents: wisesova.pitt.edu
  These anonymous websites aim to: (1) challenge negative health beliefs and increase depression/anxiety knowledge through daily blog posts enhanced with peer commentary; (2) promote social support through online peer interactions; and (3) encourage parent-adolescent mental health communication through same day blog posts with questions for discussion. Parents and adolescents cannot log on to each other's sites. The sites are moderated by our research team.
  The SOVA websites include articles composed by SOVA Peer Ambassadors who are adolescents and young adults who have experienced symptoms of depression or anxiety and contribute monthly articles and regular comments.
  Arms: Supporting Our Valued Adolescents (SOVA)
Other: Enhanced Usual Care — A social worker at the Center for Adolescent and Young Adult Health (CAYAH) clinic helps to facilitate referrals from the adolescent healthcare provider (AHCP) and contacts patients who do not schedule for within-CAYAH appointments.The study will send an extra email to the parent and adolescent that contains the content of the depart summary as well as a list of psychoeducational materials, how to contact the AHCP, CAYAH social worker, and crisis resources and the AHCP's treatment recommendation which are obtained from the electronic health record. Also, each individual will receive a phone call from a research assistant who will communicate the information in the email and offer to inform the social worker or AHCP of questions the patient or parent may have.

SUMMARY:
The purpose of this pilot study is to provide preliminary findings testing the Supporting Our Valued Adolescents (SOVA) intervention, two social media sites (one for adolescents, one for parents) aiming to address negative health beliefs, knowledge about depression or anxiety, parent-adolescent communication, in a moderated online peer community, with the goal of increasing adolescent use of mental health services.

DETAILED DESCRIPTION:
Although recent evidence shows integrated care models increase service use, implementing these models is resource intense. Even in primary care settings with access to services and routine screening for depression and anxiety, patient engagement is low. This can be explained by a low perceived need for services present in both adolescents and parents. Key target mechanisms which may increase service use include: (1) parents' and adolescents' health beliefs and knowledge, (2) emotional/informational support, and (3) communication about mental health with each other. The "SOVA" or "Supporting Our Valued Adolescents" intervention aims to address these key mechanisms through two moderated social media websites (one for parents, one for adolescents) which include daily blog posts, online peer to peer interactions, and discussion guides. SOVA had undergone an iterative process of design - using stakeholder-engagement and human computer interaction techniques (PCOR K12 HS 22989-1). The goal of this process was to build a usable intervention which is stakeholder-informed. Preliminary work has found that 100 adolescents/young adults with a history of depression or anxiety symptoms and parents find the SOVA websites to have good usability. The investigators will use a pilot randomized controlled trial of SOVA to refine recruitment and retention strategies, measure implementation outcomes and investigate potential mechanisms of action in depressed and/or anxious adolescents not currently engaged in treatment and their parents; and examine parent-adolescent communication factors about mental health and relationship quality in the context of a web-based intervention.

ELIGIBILITY:
Inclusion Criteria:

Adolescent:

* Ages 12-19
* AHCP identifies depressive and/or anxiety symptoms
* Scores at least 5 or greater on the PHQ-9 (depression) and/or GAD-7 (anxiety) consistent with at least mild symptoms
* AHCP recommends adolescent to initiate a new treatment episode (no treatment in past 3 months)
* Can read and write in English
* Have completed the 6th grade
* Assent (<18 y/o)/Consent to study (18 or 19 y/o)

Parent:

* Adolescent child meets inclusion/exclusion criteria and agrees to enroll in the study
* Can read and write in English
* Have completed the 6th grade
* Consent to study

Adolescent Healthcare Provider:

* Healthcare provider (physician, nurse practitioner, physician assistant) providing clinical services in the Center for Adolescent and Young Adult Health
* Consents to study

Exclusion Criteria:

-

Adolescent:

* Actively suicidal requiring crisis/hospitalization defined as: currently having suicidal thoughts and a plan AND AHCP recommends immediate crisis services and/or evaluation for hospitalization
* History of receiving a psychiatric medication and/or psychotherapy for depression and/or anxiety in the past 3 months
* No access to internet
* No active email account

Parent:

* No access to internet
* No active email account

Adolescent Healthcare Provier:

• None

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Study retention | 6 weeks
  proportion of dyads accessing 6-week to those who access baseline surveys

SECONDARY OUTCOMES:
Intervention acceptability | at study completion, an average of 1year
  interviews with adolescent healthcare providers
Health beliefs: Stigma | 6 weeks
  The Depression Stigma Scale (Griffiths 2004) measurizes stigmatizing attitudes toward depression treatment. It is a continuous measure and the total score ranges from 0-36. There are two subscales: the personal stigma subscale which totals 0-18 and the perceived stigma subscale which totals 0-18. These two are summed for the total stigma score. A higher score indicates a worse outcome.
Health Beliefs: Beliefs about Antidepressants - Resistance | 6 weeks
  The Resistance to Antidepressant Use Questionnaire (Cohane, 2008) measures an individual's resistance toward taking antidepressant medication if prescribed. It is a continuous measure and the total score ranges from 0 to 18, with a higher score indicating greater resistance.
Health Beliefs: Beliefs about Antidepressants - Meanings | 6 weeks
  The Antidepressant Meanings Scale (Cohane, 2008) measures an individual's level of negative attitudes toward taking an antidepressant medication if prescribed. It is a continuous measure and the total score ranges from 0 to 24, with a higher score indicating more negative attitudes.
Health Beliefs: Beliefs About Therapy - Adolescents | 6 weeks
  Barriers to Adolescents Seeking Help Scale (Wilson 2005/Kuhl 1997) measures perceptions about seeking treatment from a mental health provider. The total score ranges from 1 to 11, a higher score indicated greater barriers.
Health Beliefs: Beliefs About Therapy - Parents | 6 weeks
  The Parental version of the Barriers to Help Seeking Scale (Bates, 2010) measures parental perceptions about their child seeking treatment from a mental health provider. The total score ranges from 1 to 11, a higher score indicated greater barriers.
Depression Knowledge | 6 weeks
  The Depression literacy questionnaire (Gulliver 2012) measures knowledge about depression diagnosis and treatment. The total score ranges from 0-22, with a higher score indicating greater knowledge of depression.
Anxiety Knowledge | 6 weeks
  The Anxiety literacy questionnaire (Gulliver 2012) measures knowledge about depression diagnosis and treatment. The total score ranges from 0-22, with a higher score indicating greater knowledge of anxiety.
Peer emotional/informational support | 6 weeks
  The Medical Outcome Study Social Support Scale (Sherbourne, 1991) has a single subscale named the Emotional/informational subscale which measures types of social support which either provide emotional support or provide information. This subscale ranges from 0-100, with higher levels associated with greater support.
Peer social support | 6 weeks
  Actual/Observed emotional/informational support from online coding of peer and moderator comments for types of social support
Parent-Adolescent Communication Quality-Parent Form-Openness Subscale | 6 weeks
  The Parent-Adolescent Communication Scale measures two subscales of parent communication. This measure obtains this information from the parent perspective. The degree of openness subscale has 10 questions with a range from 10 through 50 - higher scores indicating more openness in communication.
Parent-Adolescent Communication Quality-Parent Form-Extent of Problems Subscale | 6 weeks
  The Parent-Adolescent Communication Scale measures two subscales of parent communication. This measure obtains this information from the parent perspective. The extent of communication problems subscale has a range from 10 through 50 - higher scores indicating greater extent of problems with communication.
Parent-Adolescent Communication Quality-Adolescent Form-Openness Subscale | 6 weeks
  The Parent-Adolescent Communication Scale measures two subscales of parent communication. This measure obtains this information from the adolescent perspective. The degree of openness subscale has 10 questions with a range from 10 through 50 - higher scores indicating more openness in communication.
Parent-Adolescent Communication Quality-Adolescent Form-Extent of Problems Subscale | 6 weeks
  The Parent-Adolescent Communication Scale measures two subscales of parent communication. This measure obtains this information from the adolescent perspective. The extent of communication problems subscale has a range from 10 through 50 - higher scores indicating greater extent of problems with communication.
Perceived Need for Treatment - Open ended question | 6 weeks
  Open-ended question about whether adolescent/child needs any mental health service
Perceived Need for Treatment - Survey Measure | 6 weeks
  The General-Practice Users Perceived-Need Inventory (McNab, 2004) will be used to measure perceived need for treatment. There is no scoring.
Actual Receipt of Mental Health Services | 6 weeks and 3 months
  Combined measure using Electronic Health Record Chart Review and parent/adolescent self-report as well as the Actual Help Seeking Questionnaire (Rickwood 2005) which does not involve scoring.
Depressive Symptoms | 6 weeks
  Patient Health Questionnaire-9 measures depression severity with a score ranging from 0 to 27, a higher score indicating greater severity.
Anxiety Symptoms | 6 weeks
  Generalized Anxiety Disorders 7-item Questionnaire measures extent of anxiety symptoms. The total score ranges from 0 to 21 with a higher score indicating greater severity.
Functioning | 6 weeks
  The Multidimensional Adolescent Functioning Scale (Wardennar 2013) has 3 subscales of functioning for adolescents - in general, related to family, and related to peers. The total score subscales for general are 0-40; for family are 0-28; and for peer are 0-24 with a higher score indicating higher functioning. The subscales can be totalled for a range of 0-92.
Relationship Quality | 6 weeks
  Parent-child connectedness scale, 5 questions on a 5-point Likert scale, higher scores indicated greater connectedness
Adolescent Help Seeking - Adolescent Perception | 6 weeks
  Actual Help Seeking Questionnaire, a list of individuals help may have been sought from with indication of whether this person was seen for an emotional problem in the past 2 weeks yes or no
Adolescent Help Seeking - Parent Perception of Adolescent Help Seeking | 6 weeks
  Actual Help Seeking Questionnaire, a list of individuals help may have been sought from with indication of whether this person was seen for an emotional problem in the past 2 weeks yes or no
Parent Help Seeking (for Parent themselves) | 6 weeks
  Actual Help Seeking Questionnaire, a list of individuals help may have been sought from with indication of whether this person was seen for an emotional problem in the past 2 weeks yes or no
Parent perception of Adolescent Functioning | 6 weeks
  Columbia Impairment Scale, Parent rates on a 0-4 scale how much of a problem different aspects of adolescent functioning have been, 13 item questionnaire, higher score indicates greater problems with functioning

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Adolescent and Young Adult Health, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Radovic A, DeMand AL, Gmelin T, Stein BD, Miller E. SOVA: Design of a stakeholder informed social media website for depressed adolescents and their parents. J Technol Hum Serv. 2018;35(3):169-182. doi: 10.1080/15228835.2017.1347552. Epub 2017 Jul 24. PMID 29743822
- [Background] Radovic A, Li Y, Landsittel D, Stein BD, Miller E. A Social Media Website (Supporting Our Valued Adolescents) to Support Treatment Uptake for Adolescents With Depression and/or Anxiety and Their Parents: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2019 Jan 23;8(1):e12117. doi: 10.2196/12117. PMID 30672741
- [Background] Radovic A, Odenthal K, Flores AT, Miller E, Stein BD. Prescribing Technology to Increase Uptake of Depression Treatment in Primary Care: A Pre-implementation Focus Group Study of SOVA (Supporting Our Valued Adolescents). J Clin Psychol Med Settings. 2020 Dec;27(4):766-782. doi: 10.1007/s10880-019-09669-5. PMID 31630347
- [Derived] Radovic A, Li Y, Landsittel D, Odenthal KR, Stein BD, Miller E. A Social Media Website (Supporting Our Valued Adolescents) to Support Treatment Uptake for Adolescents With Depression or Anxiety: Pilot Randomized Controlled Trial. JMIR Ment Health. 2022 Oct 7;9(10):e35313. doi: 10.2196/35313. PMID 36206044

DOCUMENTS (1):
  • Informed Consent Form (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT03318666/ICF_000.pdf